CLINICAL TRIAL: NCT07098806
Title: A Multicenter Phase 1 Study to Determine the Safety and Efficacy of Multiple Doses at Defined Intervals of Rhenium (186Re) Obisbemeda (Rhenium-186 NanoLiposome, 186RNL) Administered Via Intraventricular Catheter for Any Primary Solid Tumor Cancer With Leptomeningeal Metastases
Brief Title: Multiple Dose Intraventricular Administration of Rhenium-186 NanoLiposome for Leptomeningeal Metastases
Acronym: CA2024-LM-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Plus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA-2024-LM-001
Record Dates: First submitted 2025-07-02; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Leptomeningeal Metastasis
Keywords: Neoplastic Processes Neoplasms; Neoplasms; Pathologic Processes; Meningeal Neoplasms; Central Nervous System Neoplasms; Nervous System Neoplasms; Neoplasms by Site; Nervous System Diseases; Neoplasm Metastasis; Meningeal Carcinomatosis
MeSH Terms: conditions — Meningeal Carcinomatosis; Neoplasms; Pathologic Processes; Meningeal Neoplasms; Central Nervous System Neoplasms; Nervous System Neoplasms; Neoplasms by Site; Nervous System Diseases; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: Multiple Doses (Experimental): This is an open-label, multicenter, Phase 1 study to determine the safety and efficacy of multiple doses at defined intervals of rhenium (186Re) obisbemeda (rhenium-186 nanoliposome, 186RNL) administered via intraventricular catheter for any primary solid tumor cancer with leptomeningeal metastases to identify an MTD/MFD for a given dose, interval duration, and number of doses.
  Interventions: Drug: 186RNL

INTERVENTIONS:
Drug: 186RNL — Multiple Doses of 186RNL

SUMMARY:
This is an open-label, multicenter, Phase 1 study to determine the safety and efficacy of multiple doses at defined intervals of rhenium (186Re) obisbemeda (rhenium-186 nanoliposome, 186RNL) administered via intraventricular catheter for any primary solid tumor cancer with leptomeningeal metastases to identify an MTD/MFD for a given dose, interval duration, and number of doses.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Ability to understand the purposes and risks of the study and has signed a written informed consent document approved by the site-specific IRB.
3. Documented LM from any primary solid tumor cancer per EANO-ESMO Clinical Practice Guidelines (Types I or IIA-C).
4. Karnofsky performance status of 70 to 100.
5. Acceptable liver function:

   1. Bilirubin ≤ 1.5 times the upper limit of normal.
   2. AST (SGOT) and ALT (SGPT) ≤ 3.0 times the upper limit of normal for subjects with normal liver.
   3. AST (SGOT) and ALT (SGPT) ≤ 5.0 times the upper limit of normal for subjects with liver metastasis.
6. Acceptable renal function:

   a. Creatinine clearance greater than or equal to 60 mL/min (using the Cockcroft-Gault Equation).
7. Acceptable hematologic functioning (without hematologic support):

   1. ANC ≥ 1000 cells μL.
   2. Platelet count ≥ 75,000/μL.
   3. Hemoglobin ≥ 9.0 g/dL.
8. All women of childbearing potential must have a negative serum pregnancy test at screening. Male and female subjects must agree to use effective means of contraception (for example, surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose.
9. Normal CSF flow and distribution by an accepted CSF flow study (e.g., 111Indium-DTPA or acceptable substitute) before first treatment with the study drug, based on study imaging interpretation and clinical correlation.
10. Corticosteroids are permitted as clinically indicated.

Exclusion Criteria:

1. The subject has not recovered to the current National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v5.0) Grade ≤1 from adverse events (AEs) due to antineoplastic agents, investigational drugs, or other medications that were administered prior to study, at time of study registration.

   a. Prior AEs due to alopecia, anemia, neutropenia, and lymphopenia are not required to be recovered to Grade ≤1 prior to study registration, assuming other inclusion criteria are satisfied.
2. Contraindications to the placement of an intraventricular catheter (i.e., Ommaya reservoir.)
3. Presence of or need for a Ventriculo-peritoneal or ventriculo-atrial shunt.
4. Females of childbearing potential who are pregnant, breastfeeding, or may possibly be pregnant, without a negative serum pregnancy test (see inclusion criteria).
5. Serious intercurrent illnesses, which could interfere with the planned treatment schedule.
6. Patients who had any therapeutic radiation dose to the whole brain regardless of when the radiation treatment was delivered, except:

   1. Prior radiation dose to the spinal cord and/or cauda equina is allowed if the equivalent dose in 2 Gy fractions (EQD2) was ≤ 30 Gy to the spinal cord and/or cauda equina using α/β ratio of 3 and if prior radiotherapy has been > 14 days and ≤ 6 months, or was ≤45 Gy to the spinal cord and/or cauda equina using α/β ratio of 3 and if prior radiotherapy has been > 6 months.
   2. Prior stereotactic radiosurgery (SRS) to the brain or partial brain radiotherapy is allowed if the equivalent dose in 2 Gy fractions (EQD2) was ≤ 30 Gy to brainstem and/or optic structures (optic nerves, optic chiasm) using α/β ratio of 3 and if prior radiotherapy has been > 14 days and ≤ 6 months, or was ≤ 45 Gy to the brainstem and/or optic structures (optic nerves, optic chiasm) using α/β ratio of 3 and if prior radiotherapy has been > 6 months.
7. Prior or concurrent therapy:

   a. Intrathecally delivered therapy: i. Concurrent: Concurrent intrathecal therapy. ii. Prior: Intrathecal therapy given less than 14 days before study registration.

   b. Systemically delivered therapy: i. Concurrent: Systemically delivered therapy UNLESS LM develops while on systemically delivered therapy AND the systemically delivered therapy is NOT associated with more than grade 1 myelosuppression.

   ii. Prior: Systemically delivered therapy given less than 28 days before study registration.
8. Projected survival of less than 60 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2031-10-02 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 13 months
  Evaluation of any toxicity associated with research treatment per Common Criteria for Adverse Events.
Dose Distribution of 186RNL | 13 months
  SPECT imaging of the radioactive materials spread in the Cerebrospinal Fluid.
Safety and tolerability of multiple dose treatment | 13 months
  Evaluation of any toxicity associated with research treatment as determined by National Cancer Institute (NCI) common Terminology Criteria for adverse events (CTCAE).

SECONDARY OUTCOMES:
Determine the objective response rate (ORR). | 13 months
  Determine the overall response rate (ORR) defined as the proportion of all evaluable participants achieving a response as the best overall response at the time of progression.
Determine the overall survival (OS). | 13 months
  The time from first treatment to date of death.
Characterize the dosimetry profile of 186RNL. | 13 months
  using the following equation to calculate the average radiation-absorbed dose in the CSF Volume (Eckerman and Endo 2008): D (Gy) = 7.126 (Gy.g/mCi.h) × A cummu. (mCi.h)/ m (g) D is the average radiation-absorbed dose in Gy. A cummu. is the cumulative radioactivity in mCi.h calculated as described above. m is the weight of the radioactivity distribution volume in grams.
  Given that there is no specific tumor mass to use for organ mass in grams identifiable post-infusion, the Sponsor proposes to use the estimated total CSF volume to calculate the absorbed dose to the CSF.
  To perform radiation-absorbed dose calculation, the weight will be calculated from the average CSF volume (Adult Male: 140 ml; Adult Female: 120 ml), assuming the density of 1 g/cm3.
Determine neurologic progression-free survival (PFS). | 13 months
  The time from first treatment to progression.
Evaluate Neurologic status by NANO scale | 13 months
  Neurologic Assessment in Neuro- Oncology (NANO) The NANO scale is a quantifiable evaluation of 9 relevant neurologic domains based on direct observation and testing conducted during routine office visits. The score defines overall response criteria. The scale scores nine domains: gait, strength, ataxia, sensibility, visual fields, facial paralysis, language, level of consciousness, and behavior. Each domain has a score between 0 and 2 or 3, with 0 indicating normal function and higher scores indicating increasing deficits.

OTHER OUTCOMES:
Exploratory: Assess response using CSF tumor cell enumeration and compare to standard of care cytology. | 13 months
  Comparing the diagnostic accuracy of CNSide (cell capture and ctDNA) with cytology in diagnosing and monitoring LM and will be described in terms of sensitivity, specificity, Positive Predictive Value (PPV) and Negative Predictive Value (NPV) (as appropriate statistically).
Exploratory: Assess response using pharmacodynamic (PD) markers. | 13 months
  Determination of DNA damage markers by regression analyses of the time-activity curves will be performed and the residence times of 186RNL in red marrow will be computed using a reduction factor of 0.3 to consider the difference in activity between blood and marrow.
Safety: Determination of the incidence and severity of adverse events (AE) and serious adverse events (SAE). | 13 months
  Safety will be evaluated by the incidence of AEs and SAEs graded according CTCAE version 5.0
Safety: Determination of the incidence of dose limiting toxicities (DLT). | 13 months
  Maximum Tolerated Dose (MTD) will be evaluated by testing increasing doses with 3 to 6 participants in each cohort. MTD reflects the highest dose of drug that did not cause a Dose Limiting Toxicity (DLT) in > 33% of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- The Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No